CLINICAL TRIAL: NCT07090941
Title: Trial of Endovascular Treatment in Acute Basilar Artery Occlusion Patients With a Large Infarct Core
Brief Title: EVT in Acute Basilar Artery Occlusion With Large Infarction Core
Acronym: BOLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Hainan Medical University (Other Government)
Responsible Party: Principal Investigator, zhaozhenqiang, Principal Investigator, The First Affiliated Hospital of Hainan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOLT
Record Dates: First submitted 2025-07-13; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Basilar Artery Occlusion; Large Ischemic Core; Large Core Infarct; Endovascular Treatments
Keywords: Basilar Artery Occlusion; Endovascular treatment; Large infarct core

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Treatment Group (Experimental): Endovascular treatment procedures will be performed in accordance with each center's standard operating protocols. Based on the characteristics of vascular lesions and clinical judgment, investigators may select appropriate interventions for stenosis or occlusion, including stent retriever thrombectomy, aspiration thrombectomy, balloon angioplasty, stenting, intra-arterial thrombolysis, or various combinations of these methods.
  Interventions: Procedure: Endovascular Treatment
- Best Medical Management Group (No Intervention): Participants receive the best medical management only. Best Medical Treatment and maximum supportive care according to local guidelines, not including mechanical thrombectomy or intra-arterial treatment.

INTERVENTIONS:
Procedure: Endovascular Treatment — The vascular access route is selected based on the patient's anatomical characteristics and operator discretion. Endovascular treatment (EVT) procedures must adhere to each participating center's standardized operating protocols. Upon confirmation of vascular occlusion, EVT may be performed using devices approved by China's National Medical Products Administration (NMPA). Based on lesion-specific features and operator judgment, permissible techniques include stent retriever thrombectomy, aspiration thrombectomy, balloon angioplasty with or without stenting, or intra-arterial thrombolysis. Investigational devices are strictly prohibited.
  Arms: Endovascular Treatment Group

SUMMARY:
A multicenter, prospective, open-label, blinded endpoint, randomized controlled trial designed to evaluate the efficacy and safety of best medical management (BMM) combined with endovascular treatment (EVT) versus BMM alone in acute basilar artery occlusion (BAO) patients with large infarct cores.

DETAILED DESCRIPTION:
This trial aims to evaluate whether best medical management (BMM) combined with endovascular treatment (EVT) versus BMM alone improves neurological outcomes in acute basilar artery occlusion (BAO) patients with large infarct cores. A centralized 1:1 simple randomization design assigns participants to receive either EVT or BMM based on randomization results.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years. 2. Symptoms and signs consistent with basilar artery ischemia. 3. Basilar artery or vertebral artery occlusion confirmed by computed tomography angiography (CTA), magnetic resonance angiography (MRA), digital subtraction angiography (DSA); if vertebral artery occlusion is present, it must completely obstruct blood flow to the basilar artery.

  4. POST-NIHSS score ≥10 at randomization. 5. Time from symptom onset to randomization ≤24 hours (symptom onset defined as last known well time).

  6. pc-ASPECTS of 3-5 on CT/MRI (for patients aged <80 years) or pc-ASPECTS of 3-7 (for patients aged ≥80 years).

  7. Willingness of the patient or legally authorized representative to comply with protocol requirements and data collection procedures, with documented informed consent.

Exclusion Criteria:

* 1. Pre-stroke modified Rankin Scale (mRS) score >2. 2. Factors in the target vessel that are expected to prevent completion of endovascular treatment.

  3. Concurrent anterior and posterior circulation strokes or multivessel occlusions.

  4. Significant mass effect with imaging or clinical signs of obstructive hydrocephalus or tonsillar herniation.

  5. Basilar artery occlusion confirmed as chronic by prior imaging or investigator judgment.

  6. Presence of untreated intracranial aneurysms, intracranial tumors (except small meningiomas), or intracranial vascular malformations.

  7. Intracranial hemorrhage within the past 6 months, including parenchymal brain hemorrhage, intraventricular hemorrhage, or subarachnoid hemorrhage.

  8. Presence of active bleeding, coagulation disorders, or uncorrectable bleeding tendencies.

  9. Severe heart, liver, or kidney dysfunction or other severe systemic late-stage diseases.

  10. Known allergy to iodine contrast agents or other treatment-related drugs. 11. Medically uncontrolled refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg) (Note: Participants can be included if their blood pressure is controllable with medication and maintained at an acceptable level).

  12. Uncontrollable blood glucose <2.8 mmol/L or >22.2 mmol/L. 13. Pregnancy or breastfeeding. 14. Life expectancy <6 months. 15. Participation in other clinical studies that may affect outcome assessment. 16. Investigator's judgment that the patient is unsuitable for participation in this study or may face significant risks (e.g., due to mental illness, cognitive, or emotional disorders preventing understanding and/or compliance with study procedures and/or follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Shift analysis of the improvement trend in modified Rankin Scale (mRS) scores at 90 (±7) days after randomization. | 90 (±7) days after procedure
  Shift analysis is a statistical method used to evaluate the overall distribution change in modified Rankin Scale (mRS) scores, assessing whether an intervention leads to a general shift toward better outcomes across all score categories.

SECONDARY OUTCOMES:
Proportion of patients with a modified Rankin Scale (mRS) score of 0-3 at 90 (±7) days after randomization. | 90 (±7)days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Proportion of patients with a modified Rankin Scale (mRS) score of 0-2 at 90 (±7) days after randomization. | 90 (±7) days after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Change in POST-NIHSS score from baseline at 24 hours postoperatively. | 24 hours after procedure
  The POST-NIHSS (Posterior National Institutes of Health Stroke Scale) is a tool used to assess the severity of stroke symptoms by evaluating various neurological functions, such as consciousness, vision, movement, and speech. The score helps in gauging the degree of impairment caused by a stroke.
Change in POST-NIHSS score from baseline at discharge or 5-7 days postoperatively. | Discharge or 5 -7 days after procedure.
  The POST-NIHSS (Posterior National Institutes of Health Stroke Scale) is a tool used to assess the severity of stroke symptoms by evaluating various neurological functions, such as consciousness, vision, movement, and speech. The score helps in gauging the degree of impairment caused by a stroke.
Successful reperfusion postoperatively. | At the end of the operation
  The eTICI (extended Thrombolysis in Cerebral Infarction) score is a standard used to evaluate the degree of reperfusion in acute ischemic stroke patients following endovascular therapy (EVT). It is a further refinement of the mTICI (modified TICI) score.

OTHER OUTCOMES:
All-cause mortality at 90 (±7) days after randomization. | 90 (±7) days after procedure
  All-cause mortality refers to the rate of death from any cause within a specific time period, without considering the underlying cause of death.
Incidence of symptomatic intracerebral hemorrhage (sICH) within 48 hours after randomization (Heidelberg bleeding classification). | Within 48 hours after procedure
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 48 hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma. The sICH was defined as ICH associated with a worsening of 4 or more points on the NIHSS or resulting in death and cerebral herniation, which were not present at baseline.
Incidence of any intracerebral hemorrhage within 48 hours after randomization (Heidelberg bleeding classification). | within 48 hours after procedure
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 48 hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes